CLINICAL TRIAL: NCT04022915
Title: PET Fibrin Imaging of DVT and PE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Caravan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Peter Caravan, Associate Professor of Radiology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018P000523
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: Subjects with acute pulmonary embolism meeting the inclusion criteria will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acute pulmonary embolism (Experimental): Subjects will receive 64Cu-FBP8 and undergo PET-CT imaging.
  Interventions: Drug: 64Cu-FBP8; Diagnostic Test: PET-CT imaging

INTERVENTIONS:
Drug: 64Cu-FBP8 — Up to 10 mCi (millicurie) 64Cu-FBP8 will be administered to each subject.
Diagnostic Test: PET-CT imaging — All subjects will undergo PET-CT imaging after administration of 64Cu-FBP8.

SUMMARY:
This study aims to investigate a novel positron emission tomography(PET)-probe for imaging of fresh intravascular blood clots in pulmonary embolism (PE) and deep venous thrombosis (DVT).

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is one of the most common causes of death in the United States, resulting in more than 100,000 deaths annually. Current diagnostic techniques rely on indirect measures of clot for diagnosis and therefore suffer from the problems of both under and overdiagnosis and cannot always be performed on patients with renal failure and lung disease. In this study, we will use the novel fibrin-specific probe 64CU-FBP8 (Copper-64 labeled fibrin binding probe 8) for PET imaging of fresh blood clots in PE and DVT. Our long-term goal is to establish a novel thrombus body scan (TBS) using 64CU-FBP8 for PET imaging to overcome the limitations of indirect venous thromboembolism diagnosis, and, with one single test, provide a total-body assessment of fresh intravascular clot.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with a clinically significant pulmonary embolus (PE) confirmed by a filling defect in CT angiography (CTA), and
* Subjects must receive the radiotracer injection within 72 hours of their diagnosis.

Exclusion Criteria:

* Subjects < 18 years of age
* Time of expected radiotracer injection > 72 hours from the time of a positive venous duplex ultrasound or CT- angiogram
* Women subjects of childbearing potential who are pregnant, seeking to become pregnant, or have a positive serum pregnancy (beta-HCG) test
* Unable to lie flat for 45 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis, dyspnea),
* Weight that exceeds the PET camera table limit (300 kg)
* The subject will not be enrolled in the study if the radiation exposure for research studies during the prior 12 months, combined with the exposure from this study would exceed 50 mSv (millisievert).
* Due to the radiation exposure from imaging studies, all women of childbearing potential will be required to have a negative serum pregnancy test performed prior to any imaging procedures on the same day (if not already done that day). Patients with a positive serum pregnancy test will be excluded. Breast feeding women will also be excluded.
* A pre-existing condition or use of a medication including vasopressors and tPA (tissue Plasminogen Activator) that in the opinion of the investigator may place the subject at a substantially increased risk
* Hemodynamic instability, including requiring escalating doses of vasopressor medication.
* No groups designated as "special vulnerable populations" will be studied.
* No exclusions will be made based on race, sex, or ethnic origin.
* 64Cu-FBP8 (Copper-64 labeled fibrin binding probe 8) is cleared by the kidneys, patients with eGFR (estimated Glomerular Filtration Rate ) < 30 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Location of the thrombus within the lungs | 4 hours
  To determine the location of the thrombus regions of interest (ROIs) within the lungs using PET-CT imaging in comparison to the ROI of filling defects on CT-angiogram.
Location of clot burden measurements within the thigh | 4 hours
  To determine the location of the thrombus ROI within the thigh using PET-CT imaging in comparison to the clot on venous duplex ultrasound.
Assessment of 64Cu-FBP8 fibrin activity in the pelvic and upper extremity | 4 hours
  The prevalence of high 64Cu-FBP8 fibrin activity in the pelvic ROI and upper extremity ROI's will be reported.

SECONDARY OUTCOMES:
Correlation between normalized 64Cu-FBP8 fibrin activity and plasma D-dimer | 4 hours
  Correlation of the total fibrin activity in the imaged fields, excluding the liver, gallbladder, kidneys and urinary bladder normalized by injected dose with the plasma D-dimer.
Overall clot burden within the lungs | 4 hours
  Overall clot burden calculated as sum of 64Cu-FBP8 activity within a thrombus ROI(s) within the lungs.
Overall clot burden within the thigh | 4 hours
  Overall clot burden calculated as sum of 64Cu-FBP8 activity within a thrombus ROI(s) within the thigh.

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Winkler, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States